CLINICAL TRIAL: NCT01213381
Title: A Phase I Study Evaluating the Safety and Pharmacokinetics of SAR240550 Administered Twice Weekly in Patients With Advanced Solid Tumors.
Brief Title: Safety and Pharmacokinetics of SAR240550 (BSI-201) Twice Weekly in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED11451; U1111-1117-3152 (Other: UTN)
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Advance Solid Tumors
MeSH Terms: interventions — iniparib; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAR240550 (Experimental): * single cohort: SAR240550
  * combination cohort: SAR240550 in combination with Gemcitabine and Carboplatin
  Interventions: Drug: Iniparib (SAR240550 - BSI-201); Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Iniparib (SAR240550 - BSI-201) — Pharmaceutical form:sterile aqueous solution
  Route of administration: intravenous
Drug: Gemcitabine — Pharmaceutical form:sterile aqueous solution
  Route of administration: intravenous
Drug: Carboplatin — Pharmaceutical form:sterile aqueous solution
  Route of administration: intravenous

SUMMARY:
Primary Objective:

- To determine a dose of SAR240550 to be further studied in combination with chemotherapy regimens

Secondary Objectives:

* To determine the dose limiting toxicity (DLT) of SAR240550 and SAR240550 in combination with chemotherapy regimen (gemcitabine and carboplatin
* To assess safety profiles: significant laboratory changes and adverse events (AEs)
* To make a preliminary assessment of antitumor effect in study subjects per Response Evaluation Criteria in Solid Tumors (RECIST) with measurable disease
* To characterize SAR240550 and metabolites, 4-iodo-3-amino benzamide (IABM) and 4-iodo-3-amino-benzoic acid (IABA), pharmacokinetics
* To collect blood samples for glutathione S-transferase (GST) genotypes at baseline)

Based on data generated by BiPar/Sanofi, it is concluded that iniparib does not possess characteristics typical of the PARP inhibitor class. The exact mechanism has not yet been fully elucidated, however based on experiments on tumor cells performed in the laboratory, iniparib is a novel investigational anti-cancer agent that induces gamma-H2AX (a marker of DNA damage) in tumor cell lines, induces cell cycle arrest in the G2/M phase in tumor cell lines, and potentiates the cell cycle effects of DNA damaging modalities in tumor cell lines. Investigations into potential targets of iniparib and its metabolites are ongoing.

DETAILED DESCRIPTION:
The duration of the study for each patient will include an up to 4-week screening phase, 21-day study cycle(s), followed by a 30 day follow-up.

ELIGIBILITY:
Inclusion criteria:

- Histologically or cytologically documented advanced solid tumor that was refractory to standard therapy or for which no standard therapy is available

Exclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of ≥2
* Known hematological malignancies
* Symptomatic or untreated brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation, and corticosteroids
* Myocardial infarction within 6 months of study Day 1, unstable angina, congestive heart failure with New York Heart Association >class II, uncontrolled hypertension
* Active human immunodeficiency virus infection, hepatitis C virus, or chronic hepatitis B infection
* Major surgery within 28 days of study Day 1
* Not recovered from all previous therapies (i.e. radiation, surgery, and medications)
* Adverse events related to previous therapies must be Common Terminology Criteria for Adverse Events (CTCAE) grade ≤ 1 (except alopecia) at screening or returned to the subject's baseline prior to their most recent previous therapy
* Inadequate organ and bone marrow function Radiation therapy within 14 days of study Day 1
* Chemotherapy or antibody therapy for treatment of underlying malignancy within 21 days of study Day 1
* Concurrent or prior (within 7 days of study Day 1) anticoagulation therapy
* Currently enrolled or was enrolled within 30 days of completing other investigational drug study, or receiving other investigational agent not approved for any indications
* Subject who had been previously enrolled in this study . Not available for follow-up assessment
* Any kind of disorder that compromised the ability of the subject to give written informed consent and/or comply with the study procedures
* Patient who is judged by the investigator as not suitable for participation in the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity in cycle 1 | 3 Weeks

SECONDARY OUTCOMES:
Efficacy assessment as tumor response defined by Response Evaluation Criteria in Solid Tumors (RECIST) | 30 days after the last injection
Safety based on clinical and laboratory tests and Adverse Events (AEs) | 30 days after the last injection
Pharmacokinetics of SAR240550 | Cycle 1 and Cycle 2
Pharmacodynamics of SAR240550 | Cycle1, Cycle 2 and 30 days after the last injection
Pharmacogenomic analysis of glutathione S-transferase (GST) genotypes | Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Japan (2):
  - Sanofi-Aventis Investigational Site Number 392001, Kobe
  - Sanofi-Aventis Investigational Site Number 392002, Matsuyama